CLINICAL TRIAL: NCT01125904
Title: A Study In Trained Taste Panel Healthy Adult Volunteers To Investigate The Palatability Of Select Formulations Of Crizotinib Oral Liquid
Brief Title: A Study To Investigate The Taste Of Crizotinib Liquid In Trained Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A8081018
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Crizotinib
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib (Experimental)
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — Oral liquid. Taste assessment of new formulation. Subjects will not ingest the drug.

SUMMARY:
An oral-liquid, pediatric form of crizotinib designed for use by pediatric patients is being tested for its' palatability in adults.

DETAILED DESCRIPTION:
Taste assessment of new formulation. Subjects will not ingest the drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non childbearing potential subjects between the ages of 18 and 75 years, inclusive.
* Subjects must be trained sensory panelists.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, product evaluations, laboratory tests, and other study procedures.

Exclusion Criteria:

* A history of clinically significant hematological, renal, endocrine, pulmonary , glaucoma, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic disease (excluding untreated, asymptomatic seasonal allergies at the time of product evaluation) as evaluated through a medical history.
* A history of hypersensitivity to any inactive ingredients employed in the formulation(s).
* Receiving treatment with an investigational drug within 28 days preceding any of the product evaluations for this study.
* Participation in a product taste evaluation (ie, 'sip and spit' type taste evaluation) involving an active pharmaceutical ingredient (API) within 5 half lives of that API.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
A complete description of the sensory attributes of drug product prototype formulations (eg, aroma, flavor, texture, and mouthfeel). | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Woburn, Massachusetts, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081018&StudyName=A%20Study%20To%20Investigate%20The%20Taste%20Of%20Crizotinib%20Liquid%20In%20Trained%20Healthy%20Adult%20Volunteers%20